CLINICAL TRIAL: NCT06703385
Title: Effect of Suboccipital Release Versus Instrument- Assisted Soft Tissue Mobilization on Tension Type Headache
Brief Title: Suboccipital Release Versus Instrument- Assisted Soft Tissue Mobilization on Tension Type Headache
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nada Gamal Saad, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nada-005491
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Suboccipital Release; Instrumental Assisted Soft Tissue Mobilization; Tension-Type Headache
MeSH Terms: conditions — Tension-Type Headache

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional program (Active Comparator): Twenty patients will receive conventional physical therapy including Hot pack and exercise therapy program (ROM exercise, stretching exercise, isometric strengthening exercise for cervical muscles
  Interventions: Other: conventional physical therapy program
- suboccipital release (Experimental): Twenty patients will receive suboccipital release plus the Same conventional physical therapy program.
  Interventions: Other: Suboccipital release; Other: conventional physical therapy program
- instrumental assisted soft tissue mobilization (Experimental): Twenty patients will receive instrumental assisted soft tissue mobilization plus the Sam conventional physical therapy program.
  Interventions: Other: Instrument Assisted soft tissue mobilization; Other: conventional physical therapy program

INTERVENTIONS:
Other: Instrument Assisted soft tissue mobilization — The blade is a surgical instrument for soft tissue mobilization, made of 100% surgical stainless steel with 8 treatment planes and 2 treatment edges. It is used to locate muscle limitations and apply gentle strokes along the affected muscle, detecting changes in soft tissue consistency. The procedure is repeated three times a week for four weeks.
  Arms: instrumental assisted soft tissue mobilization
Other: Suboccipital release — The patient will lie in a relaxed supine position, with a therapist sitting on a chair. The therapist will apply pressure to the C2 area, holding it until a melting sensation is felt. The intervention time is 4 minutes. The patient will close both eyes during the Suboccipital release procedure to prevent eye movements affecting muscle tone. Interventions will be three times a week for four weeks.
  Arms: suboccipital release
Other: conventional physical therapy program — The patient is placed in a sitting position and a hot pack is applied to the back of the neck for 15 minutes. The therapist then performs active range of motion exercises for neck flexion, extension, rotation, and lateral flexion without resistance. They also perform stretching exercises for upper Trapezius muscle and suboccipital muscle. Strengthening exercises for neck muscles are performed through isometric exercises, such as side pending to right, side pending to left, extension, and flexion. The interventions are conducted three times, peer-wise, for four weeks. The treatment aims to improve neck flexibility and overall well-being.

SUMMARY:
The study aims to explore the impact of suboccipital release versus instrument-assisted soft tissue mobilization on pain intensity, pressure pain threshold, headache impact test, and headache frequency in patients with tension headache. The research will also examine the effects of these methods on headache impact tests and frequency.

DETAILED DESCRIPTION:
Headache prevalence ranges from 38.2 to 59.4%, with a lifetime prevalence of 26.1-45%. Tension Type Headache can be episodic or chronic, with 78% occurring less than 15 times/month and 6% occurring more than 15 times/month. Tension Type Headache has a greater socioeconomic burden, leading to lower productivity and workday loss. Tension Type Headache is linked to myofascial pain and trigger points, which can cause sensory changes and reduced pain threshold. Studies show that referred pain from myofascial trigger points reproduces headache in patients with , leading to increased symptom severity. Frequent Episodic tension type headache increases the risk of developing chronic tension type headache due to analgesic overuse. instrumental assisted soft tissue mobilization, a physical therapy technique, promotes fascia realignment and reduces strain on the clinician's hands.

ELIGIBILITY:
Inclusion Criteria:

1. Participants of both gender will be between the ages of 18 and 60.
2. Episodic tension type headache criteria, according to the International Headache Society's Headache Classification Committee., have at least two of the following characteristics.

   * Recurrent episodes of headache on less than 15 days per month for at least 3 months
   * Headache that last for from around 30 min till seven days.
   * At least 2 of the following features are found in a headache:
   * A location that is on two sides.
   * Tightening/pressing quality (non-pulsating).
   * Intensity is mild to moderate.
   * Both of the following: Not worsened by routine physical activity, there is no nausea or vomiting.
   * Only have one photophobia/ phonophobia
3. Patients have active trigger points in suboccipital muscle and upper trapezius muscle
4. The presence of myofascial trigger points was determined by therapist using the diagnostic criteria described by Simons .,(1999) ,The major criteria of active myofascial trigger points were: Regional neck pain, Pain or altered sensation in the expected distribution of referred pain from a myofascial trigger point, Taut band palpable in an accessible muscle.

Exclusion Criteria:

1. Patients who have had a history of cancer
2. Patients who have had cervical and cranial surgery
3. Patients with severe psychological disorders (major Depression)
4. Patients with uncontrolled hypertension
5. Dysfunctions in the tempo-mandibular joint
6. Headaches associated with high fever, stiff neck, or rash, problems of vision or profound dizziness
7. Female who are pregnant or lactating

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
assessment of pain intensity using numeric pain rating scale | at baseline and after 4 weeks
  Assessment of pain intensity using Numerical pain Rating Scale An 1l-point numeric scale with 0 representing one pain extreme(e.g., "no pain") and 10 representing the other pain extreme (e.g., "pain as bad as you can imagine" and "worst pain imaginable)

SECONDARY OUTCOMES:
Assessment of pressure pain threshold using pressure algometer | at baseline and after 4 weeks
  The Pain Pressure Threshold is measured using a pressure algometer on trapezius and suboccipital trigger points. The patient's maximum pain tolerance is recorded, and the procedure is repeated three times to calculate the average.
Assessment of the impact of headache using the Headache Impact Test questionnaire | at baseline and after 4 weeks
  The Headache Impact Test (HIT-6) is a questionnaire measuring the impact of headaches on daily activities. It consists of six questions, each scoring 6-13, with a final score ranging from 36 to 78. A higher score indicates more headache-related disability. The test categorizes headache impact severity into four categories: little or no impact (49 or less), some impact (50-55), substantial impact (56-59), and severe impact (60-78).
Assessment of Frequency of headache | at baseline and after 4 weeks
  The number of headache days per week will be used to identify it. The participant keep count of how many days they have a headache in the week previous treatment and after four weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- out-patient clinic, national institute of neuromotor system, Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No